CLINICAL TRIAL: NCT01162694
Title: Protocol: Comparing the Effect of Using an Internet-Based Glucose Monitoring System Versus the Continuous Glucose Monitoring System on HbA1c Levels in Type 2 DM
Brief Title: Comparing Internet Blood Glucose Monitoring System and Continuous Glucose Monitoring System
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was expanded and included in another study.
Sponsor: Endocrine Research Society (Other)
Responsible Party: Principal Investigator, Dr. Hugh Tildesley, Clinical Professor, Endocrine Research Society
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IBGMS vs CGMS
Record Dates: First submitted 2010-06-04; First posted 2010-07-15 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Remote Blood Glucose Monitoring System,; Continuous Glucose Monitoring System,; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Internet Intervention (Active Comparator): The subjects enrolled in the Internet Therapeutic Intervention arm receive standard care by testing their blood glucose at least 3 times daily and visit the endocrinologist every 3 months; however, they are also asked to upload their blood glucose readings online every 2 weeks for the health practitioner to view and comment upon.
  Interventions: Other: Remote Blood Glucose Monitoring
- Continuous Glucose Monitoring (Active Comparator): The use of CGMS (Sensor, receiver, transmitter) plus the uploading of results to the Internet-based software utility of CareLink Personal and generating reports that can be viewed and used at the patient's own preference. This group will send the uploaded data and receive feedback from their endocrinologist every 2 weeks.
  Interventions: Other: Continuous Glucose Monitoring

INTERVENTIONS:
Other: Remote Blood Glucose Monitoring — The subjects enrolled in the Internet Therapeutic Intervention arm receive standard care by testing their blood glucose at least 3 times daily and visit the endocrinologist every 3 months; however, they are also asked to upload their blood glucose readings online every 2 weeks for the health practitioner to view and comment upon.
  Other Names: Internet Blood Glucose Monitoring System
  Arms: Internet Intervention
Other: Continuous Glucose Monitoring — The use of CGMS (Sensor, receiver, transmitter) (Medtronic Diabetes) plus the uploading of results to the Internet-based software utility of CareLink Personal and generating reports that can be viewed and used at the patient's own preference. This group will not receive feedback or suggestion based on the uploaded glucose data.
  Other Names: Sensors, CGMS
  Arms: Continuous Glucose Monitoring

SUMMARY:
Management of type 2 diabetes is an ongoing challenge for patients and their doctors. In order to prevent short and long term complications, patients need to monitor and control their blood sugar levels. In addition, they may need to have an ongoing communication with their doctor in order to modify treatment. In this study the investigators wish to compare two systems of monitoring and communication of blood sugar levels. The first is the use of continuous glucose monitoring system and the second is the use of an Internet-based glucose monitoring system. The investigators want to compare their effect and/or benefits.

DETAILED DESCRIPTION:
Purpose: To compare the benefits of the Internet-based glucose monitoring system with the Continuous Glucose monitoring system in patients with type 2 diabetes mellitus.

Hypothesis:The investigators propose that the benefits from the Internet-based glucose monitoring system (IBGMS) will be comparable to the benefits of the Continuous Glucose monitoring system (CGMS) for patients with type 2 DM.

Justification: Half of the subject will be on the standard treatment, which will involve glucose monitoring by testing blood glucose 3 times daily, performing a laboratory test of blood hemoglobin every three months, and visiting the doctor every three months for standard care. They will also use the internet system to report their glucose readings,which will allow the health care professions to view the results and provide feedback. The other half will use the continuous glucose monitoring system, which will involve a minimum of testing blood glucose at least 2 times a day to calibrate the sensor, performing laboratory test of blood hemoglobin every three months, and visiting the doctor every three months for standard care. All of the subjects will be under standard care;

Research Method: Type 2 diabetes patients who satisfy the inclusion criteria will be recruited from St. Paul's Diabetes Teaching and Training Centre. They will be randomized into 2 groups (IBGMS and CGMS). There is an equal chance, a 50/50 chance, of being placed in either group.

The IBGMS group will receive standard care and will be asked to perform self-blood glucose monitoring 3 times daily for 6 months. The IBGMS group will also be asked to report their blood glucose reading every 2 weeks through an Internet based glucose monitoring system. The IBGMS group will make visits to the endocrinologist every 3 months with A1c and serum creatinine measurements at 3-month intervals for 6 months.

The CGMS group will also receive standard care and will be asked to perform self-blood glucose monitoring at least 2 times a day for 6 months to calibrate the sensor.The CGMS group will also be using the internet system to generate a report of their blood glucose readings and can be used at the patient's own preference. Their readings will also be sent to the endocrinologist for feedback every 2 weeks. The CGMS group will make visits to the endocrinologist every 3 months with A1c and serum creatinine measurements at 3-month intervals for 6 months. The laboratory measurements of both groups will be recorded and used for data analysis.

Statistical Analysis: The primary endpoint is the A1c level or the change in A1c level. The secondary endpoints include severe hypoglycemia defined as requiring external aid, hospital admissions for any CVD related intervention, and adverse events such as unplanned hospitalizations for any cause that last more than 24 hours. Patients who do not have the required number of SMBG (Self monitored blood glucose) tests performed or patients requiring new laser therapy will be asked to discontinue the study.

For each group, A1C levels before the start of study will be compared to A1C levels 3 and 6 months after the start of the study. Paired t-tests and random effects models (longitudinal analyses) will examine differences in A1C values before and after the study duration. Unpaired, independent t-tests will be done to examine the difference in A1C values between the two groups before and after the interventions. The planned sample size is 50.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes patients being treated with insulin for at least 3 months
* HbA1c > 7%
* > 25 years of age
* Willingness to test blood glucose levels a minimum of 3 times daily
* Willingness to be trained on using the Continuous Glucose Monitoring System
* Willingness to be randomized
* Trained in self-blood glucose monitoring
* Internet Access on a Windows Personal Computer
* No prior use or training on CGMS in the past 6 months
* No prior use or training on IBGMS in the past 6 months

Exclusion Criteria:

Patients who do not meet the above criteria or are not willing to participate will not be included in the study. Additional exclusion criteria include:

* Patient with medical conditions that may affect their study participation or results will be excluded.
* Patients with the potential to become pregnant
* Patients using medications known to influence control of diabetes (eg steroids systemic or inhaled)
* Liver disease (AST or ALT levels > 2.5 times the reference level)
* Renal insufficient with a serum creatinine level > 200 μmol/L

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the A1c level or the change in A1c level | 6 Months

SECONDARY OUTCOMES:
The secondary endpoint include severe hypoglycemia defined as requiring external aid (hospital or other). | 6 Months
A secondary endpoint includes adverse events such as unplanned hospitalizations for any cause that last more than 24 hours | 6 monthns

CONTACTS AND LOCATIONS:
Overall Officials: Hugh D Tildesley, MD, Principal Investigator — Providence Health Care, University of British Columbia
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Nathan DM, Cleary PA, Backlund JY, Genuth SM, Lachin JM, Orchard TJ, Raskin P, Zinman B; Diabetes Control and Complications Trial/Epidemiology of Diabetes Interventions and Complications (DCCT/EDIC) Study Research Group. Intensive diabetes treatment and cardiovascular disease in patients with type 1 diabetes. N Engl J Med. 2005 Dec 22;353(25):2643-53. doi: 10.1056/NEJMoa052187. PMID 16371630
- [Background] Intensive blood-glucose control with sulphonylureas or insulin compared with conventional treatment and risk of complications in patients with type 2 diabetes (UKPDS 33). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998 Sep 12;352(9131):837-53. PMID 9742976
- [Background] Hirsch IB, Bode BW, Childs BP, Close KL, Fisher WA, Gavin JR, Ginsberg BH, Raine CH, Verderese CA. Self-Monitoring of Blood Glucose (SMBG) in insulin- and non-insulin-using adults with diabetes: consensus recommendations for improving SMBG accuracy, utilization, and research. Diabetes Technol Ther. 2008 Dec;10(6):419-39. doi: 10.1089/dia.2008.0104. PMID 18937550
- [Background] Klonoff DC, Bergenstal R, Blonde L, Boren SA, Church TS, Gaffaney J, Jovanovic L, Kendall DM, Kollman C, Kovatchev BP, Leippert C, Owens DR, Polonsky WH, Reach G, Renard E, Riddell MC, Rubin RR, Schnell O, Siminiero LM, Vigersky RA, Wilson DM, Wollitzer AO. Consensus report of the coalition for clinical research-self-monitoring of blood glucose. J Diabetes Sci Technol. 2008 Nov;2(6):1030-53. doi: 10.1177/193229680800200612. PMID 19885292
- [Background] Austin MM, Haas L, Johnson T, Parkin CG, Parkin CL, Spollett G, Volpone MT. Self-monitoring of blood glucose: benefits and utilization. Diabetes Educ. 2006 Nov-Dec;32(6):835-6, 844-7. doi: 10.1177/0145721706295873. No abstract available. PMID 17102152
- [Background] Yoo HJ, An HG, Park SY, Ryu OH, Kim HY, Seo JA, Hong EG, Shin DH, Kim YH, Kim SG, Choi KM, Park IB, Yu JM, Baik SH. Use of a real time continuous glucose monitoring system as a motivational device for poorly controlled type 2 diabetes. Diabetes Res Clin Pract. 2008 Oct;82(1):73-9. doi: 10.1016/j.diabres.2008.06.015. Epub 2008 Aug 12. PMID 18701183